CLINICAL TRIAL: NCT06200714
Title: Observational, Multicentre, Prospective, Real-world Post-authorization Safety Study Describing the Achievement of Nintedanib-associated DIArrhoea Control After 12 Weeks of Follow-up in Patients With Idiopathic puLmonary FIBrosis (IPF) and Progressive Pulmonary Fibrosis (Other Than IPF) in Spain: the DIALFIB Study
Brief Title: A Study Based on Medical Records in Spain That Looks at Diarrhoea Control in People With Pulmonary Fibrosis Who Are Taking Nintedanib
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0545
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Diarrhoea
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPF patients: Clinical management of interstitial lung diseases (IPF) or other progressive pulmonary fibrosis (PPF) patients who experienced nintedanib-associated diarrhoea

SUMMARY:
This is an observational, non-interventional, and prospective post authorization safety study (PASS) that will describe the real-world proportion of patients that achieve nintedanib-associated diarrhoea control after 12 weeks of follow-up, in hospital settings in Spain. It will include outpatients (i.e., those attending ambulatory visits) with interstitial lung diseases (IPF) and other progressive pulmonary fibrosis (PPF) treated with nintedanib (150 mg bid) and having a first episode of diarrhoea after nintedanib initiation.

ELIGIBILITY:
Inclusion criteria/definition

* Adults (≥18 years old) at diarrhoea initiation.
* Ability to consent and to conduct all procedures of the study, as judged by the study investigator, and agreeing to participate providing informed consent at baseline.
* Diagnosis of idiopathic pulmonary fibrosis (IPF) or progressive pulmonary fibrosis (PPF) (other than IPF), as registered in electronic medical records (EMR) using free text or international statistical classification of diseases and related health problems (ICD) codes (ICD-9 and/or ICD-10), at least 1 day before diarrhoea initiation.
* Being treated with 150 milligram (mg) bid of nintedanib when initiating diarrhoea symptoms, defined as having a nintedanib anatomical therapeutic chemical (ATC) code (L01EX09) or the molecule/commercial name registered in the EMR, for at least 1 day before diarrhoea initiation.
* First pulmonologist consultation (face-to-face) at the time of recruitment due to a first diarrhoea episode as defined by the pulmonologist since nintedanib initiation. Diarrhoea defined as the passage of three or more loose or liquid stools in a 24-hour period (loose or liquid stools defined as stools with a Bristol Stool Form Scale (BSFS) of 6 or 7 points).

Exclusion criteria

1. Patients diagnosed with systemic sclerosis associated interstitial lung disease (SSc-ILD) as registered in EMR using free text or ICD codes (ICD-9 and ICD-10). Referent to any time before or at diarrhoea initiation.
2. Participation in any clinical trial including a drug or device at any time before or at diarrhoea initiation.
3. Participation in any Patient Support Programme (PSP) at diarrhoea initiation.
4. Having history of chronic gastrointestinal disorder (e.g., inflammatory bowel disease or the short gut syndrome), pancreatic dysfunction/insufficiency, or colon cancer; due to the likelihood of faecal incontinence. Referent to any time before or at diarrhoea initiation.
5. Having a performance status (PS) ≥3 points on the Eastern Cooperative Oncology Group scale (ECOG) scale at diarrhoea initiation, due to the likelihood of faecal incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical management of interstitial lung diseases (IPF) or other progressive pulmonary fibrosis (PPF) patients who experienced nintedanib-associated diarrhoea.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Achievement of diarrhoea control (yes/no) | Up to 12 weeks
  Achievement of diarrhoea control (yes/no), defined as the passage of less than 3 loose or liquid stools in a 24-hour period (loose or liquid stools defined as stools with a Bristol Stool Form Scale (BSFS) of 6 or 7 points while being treated with 150 mg bid of nintedanib, at 12-week follow-up.

SECONDARY OUTCOMES:
Absolute change in the proportion of patients taking optimal nintedanib dose (150 mg bid) at 12- week follow-up referent to diarrhoea initiation | Up to 12 weeks
Absolute change in Bristol Stool Form Scale (BSFS) score at week 12 follow-up referent to diarrhoea initiation | Up to 12 weeks
Absolute change in number of stools per day at 12- week follow-up referent to diarrhoea initiation | Up to 12 weeks
Absolute change in current body weight (in kilograms) at 12-week follow-up referent to diarrhoea initiation | Up to 12 weeks
Proportion of patients using carob flour for the treatment of nintedanib-associated diarrhoea at any time from diarrhoea initiation to 12-week follow-up | Up to 12 weeks
Number of patients per treatment category for nintedanib-associated diarrhoea at diarrhoea initiation | Up to 12 weeks
  Treatment categories of nintedanib-associated diarrhoea could include pharmacological treatments (e.g., loperamide) or non-pharmacological treatment (e.g., carob flour, zinc, probiotics, other dietary interventions, hydration)
Number of patients per treatment category for nintedanib-associated diarrhoea at 12-week follow-up | Up to 12 weeks
  Treatment categories of nintedanib-associated diarrhoea could include harmacological treatments (e.g., loperamide) or non-pharmacological treatment (e.g., carob flour, zinc, probiotics, other dietary interventions, hydration).
Occurrence of at least one dose reduction (yes/no), defined as reduction of nintedanib dose from 150 mg bid to 100 mg bid, from diarrhoea initiation to 12-week follow-up | Up to 12 weeks
Occurrence of permanent withdrawal, defined as discontinuing 150 mg bid or 100 mg bid of nintedanib and not reintroducing it before the 12- week follow-up) | Up to 12 weeks
Occurrence of at least one dose escalation (yes/no), defined as an increase of nintedanib dose from 100 mg bid to 150 mg bid from diarrhoea initiation to 12-week follow-up | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario de Cruces, Bizkaia
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital de La Princesa, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Álvaro Cunqueiro, Pontevedra
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame frame' are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents upon signing of a 'Document Sharing Agreement'. For study data 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com